CLINICAL TRIAL: NCT04854057
Title: Combinatorial Treatment of Acute Intermittent Hypoxia and Transcutaneous Electrical Spinal Cord Stimulation to Improve Hand Function in People With Cervical Spinal Cord Injury
Brief Title: Pairing Intermittent Hypoxia and Transcutaneous Electrical Spinal Cord Stimulation to Promote Arm Use After Cervical SCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding or personnel for project. We are unable to meet the recruitment goals for this pilot study.
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Randy Trumbower, PT, PhD, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P003328
Record Dates: First submitted 2021-04-14; First posted 2021-04-22 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injuries
Keywords: hypoxia; spinal cord injury; rehabilitation; function; low oxygen
MeSH Terms: conditions — Spinal Cord Injuries; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First (Experimental): Round 1 1st Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 1 2nd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Round 1 3rd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Washout (1 month)
  Round 2 1st Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 2 2nd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM.
  Round 2 3rd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH.
  Interventions: Other: AIH - Intermittent Hypoxia - hypoxia air mixture; Other: SHAM - Intermittent Room Air - room air mixture; Device: TESS - Transcutaneous Electrical Spinal Cord Stimulation + Functional Task Practice
- Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First (Experimental): Round 1 1st Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 1 2nd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM.
  Round 1 3rd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH.
  Washout (1 month)
  Round 2 1st Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 2 2nd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Round 2 3rd Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Interventions: Other: AIH - Intermittent Hypoxia - hypoxia air mixture; Other: SHAM - Intermittent Room Air - room air mixture; Device: TESS - Transcutaneous Electrical Spinal Cord Stimulation + Functional Task Practice

INTERVENTIONS:
Other: AIH - Intermittent Hypoxia - hypoxia air mixture — Participants will breathe intermittent low oxygen via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of fraction of inspired oxygen (FIO2)=0.10±0.02 (hypoxia). Participants will receive treatment 4 times per week.
Other: SHAM - Intermittent Room Air - room air mixture — Participants will breathe intermittent room air via air generators. The generators will fill reservoir bags attached to a non-rebreathing face mask. Oxygen concentration will be continuously monitored to ensure delivery of fraction of inspired oxygen (FIO2)=0.21±0.02 (normoxia). Participants will receive treatment 4 times per week.
Device: TESS - Transcutaneous Electrical Spinal Cord Stimulation + Functional Task Practice — Participants will receive transcutaneous electrical stimulation to the cervical spinal cord using the TESCoN device developed by SpineX, Inc. Training will consist of progressive functional task practice for upper extremity motor training. A total of 24 treatment sessions, which will last 45 minutes per session, will be completed in 3 weeks (4 days/week) per crossover arm.

SUMMARY:
The purpose of this study is to test the efficacy of mild breathing bouts of low oxygen (intermittent hypoxia) combined with transcutaneous electrical spinal cord stimulation on restoring hand function in persons with chronic incomplete spinal cord injury.

DETAILED DESCRIPTION:
The goal of this study is to determine the effectiveness of repeatedly breathing mild bouts of low oxygen for brief periods (termed acute intermittent hypoxia (AIH)) combined with non-invasive transcutaneous electrical spinal cord stimulation (TESS) on restoring hand function in persons with chronic incomplete SCI.

The fundamental hypothesis guiding this proposal is that daily AIH+TESS engage excitatory and inhibitory pathways, which converge on a common plasticity-promoting cascade that induces greater recovery of hand function than either one alone.

Both treatments appear to enhance motor function in persons with cervical SCI. Despite their independent effects on promoting functional benefits, it is not yet know if they may promote greater functional benefits when combined. To be effective as a long-term rehabilitation strategy, it is essential to determine the efficacy of combined protocols of recurring AIH+TESS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* medically stable with medical clearance from physician to participate
* SCI at or below C3 and at or above C7
* non-progressive etiology of spinal injury
* American Spinal Injury Association Impairment Scale (AIS) C-D at initial screen
* at least 1 year post-injury (chronic)
* difficulty independently performing hand functions in activities of daily living

Exclusion Criteria:

* dependence on ventilation support
* implanted stimulator (e.g. diaphragm pacing by phrenic nerve stimulation, vagus nerve stimulator, pacemaker, cochlear implant, epidural stimulator, baclofen pump, etc.)
* spinal cord injury related complications including unhealed pressure sore, severe neuropathic or chronic pain syndrome, history of frequent autonomic dysreflexia, infection (e.g. urinary tract), cardiovascular disease (e.g. deep vein thrombosis), pulmonary disease, heterotopic ossification in the upper extremities, severe osteoporosis, unhealed fracture, contracture of the upper extremity joints
* received botulinum toxin injections in upper extremity muscles in the prior 6 months
* history of tendon or nerve transfer surgery in the upper extremity
* history of additional neurologic disease, such as stroke, multiple sclerosis, traumatic brain injury, peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.) or peripheral nerve injury in the upper extremity
* history of concomitant diseases that would prevent full participation in intensive exercise therapy, such as uncontrolled hypertension, rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.), pulmonary disease, active cancer, chronic contagious disease, etc.
* anticoagulation medication
* pregnancy
* history of allergic reaction or any skin reaction to use of adhesive electrodes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Trumbower, PT, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Trumbower RD, Hayes HB, Mitchell GS, Wolf SL, Stahl VA. Effects of acute intermittent hypoxia on hand use after spinal cord trauma: A preliminary study. Neurology. 2017 Oct 31;89(18):1904-1907. doi: 10.1212/WNL.0000000000004596. Epub 2017 Sep 29. PMID 28972191
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Hoffman L, Field-Fote E. Effects of practice combined with somatosensory or motor stimulation on hand function in persons with spinal cord injury. Top Spinal Cord Inj Rehabil. 2013 Fall;19(4):288-99. doi: 10.1310/sci1904-288. PMID 24244094
- [Background] Gad P, Lee S, Terrafranca N, Zhong H, Turner A, Gerasimenko Y, Edgerton VR. Non-Invasive Activation of Cervical Spinal Networks after Severe Paralysis. J Neurotrauma. 2018 Sep 15;35(18):2145-2158. doi: 10.1089/neu.2017.5461. PMID 29649928
- See also: INSPIRE Lab - dedicated to inspire persons with paralysis to move again — https://www.inspire-lab.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First: Round 1 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 1 Second Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Round 1 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Washout (1 month)
  Round 2 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 2 Second Intervention (4 days):Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Round 2 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
- Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First: Round 1 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 1 Second Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Round 1 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Washout (1 month)
  Round 2 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 2 Second Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Round 2 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
Period: Overall Study
Arm/Group | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3
Upper Extremity Function [Mean (Full Range); unit: units on a scale] — Upper extremity function performance metrics assessed using the Graded Redefined Assessment of Strength, Sensation and Prehension test (GRASSP v2). Range: 0 to 188. Higher values represent a better outcome.
  units on a scale
    Round 1 | 39 [39 to 39] | 91 [27 to 155] | 74.7 [27 to 155]
    Round 2 | 47 [47 to 47] | 90.5 [22 to 159] | 76 [22 to 159]
Upper Extremity Strength - Cylindrical Grip - Less Impaired Hand [Mean (Full Range); unit: kg] — Upper extremity strength assessed using dynamometers to measure grip forces.
  kg
    Round 1 Baseline | 3.5 [3.5 to 3.5] | 14.3 [.5 to 28.1] | 10.7 [.5 to 28.1]
    Round 2 Baseline | 3.6 [3.6 to 3.6] | 17.45 [.9 to 34.0] | 12.8 [.9 to 34.0]
Upper Extremity Strength - Cylindrical Grip - More Impaired Hand [Mean (Full Range); unit: kg] — Upper extremity strength assessed using dynamometers to measure grip forces.
  kg
    Round 1 Baseline | 0 [0 to 0] | 12.7 [0 to 25.4] | 8.5 [0 to 25.4]
    Round 2 Baseline | 0 [0 to 0] | 15.1 [0 to 30.1] | 10.0 [0 to 30.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Function
Description: Change compared to baseline in upper extremity function performance metrics after treatment assessed using the Graded Redefined Assessment of Strength, Sensation and Prehension test (GRASSP v2). Range: -188 to 188. Higher values represent a better outcome.
Time Frame: Once each intervention week (days 5, 10, and 15), and once at follow-up (week 8)
Population: 1 subject from SHAM+TESS First group dropped out after round 2 day 5.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First
Number analyzed (Participants) | 1 | 2
score on a scale
  Round 1 Day 5 | -2 [-2 to -2] | 6 [-1 to 13]
  Round 1Day 10 | 5 [5 to 5] | 7 [-1 to 15]
  Round 1 Day 15 | 6 [6 to 6] | 7 [-3 to 17]
  Round 1 Week 8 | 8 [8 to 8] | -0.5 [-5 to 4]
  Round 2 Day 5 | -1 [-1 to -1] | 11.5 [6 to 17]
  Round 2 Day 10: number analyzed (Participants) | 1 | 1
  Round 2 Day 10 | 1 [1 to 1] | 18 [18 to 18]
  Round 2 Day 15: number analyzed (Participants) | 1 | 1
  Round 2 Day 15 | -2 [-2 to -2] | 17 [17 to 17]
  Round 2 Week 8: number analyzed (Participants) | 1 | 1
  Round 2 Week 8 | 0 [0 to 0] | 16 [16 to 16]

2. Primary Outcome: Change in Upper Extremity Strength - Cylindrical Grip - Less Impaired Hand
Description: Change in upper extremity strength compared to baseline assessed using dynamometers to measure grip forces.
Time Frame: Once each intervention week (days 5, 10, and 15), and once at followup (week 8)
Population: 1 subject from SHAM+TESS First group dropped out after round 2 day 5.
Measure: Mean (Full Range); unit: kg
Arm/Group | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First
Number analyzed (Participants) | 1 | 2
kg
  Round 1 Day 5 | -.47 [-.47 to -.47] | 1.65 [0 to 3.30]
  Round 1 Day 10 | -.63 [-.63 to -.63] | 1.63 [-0.33 to 3.60]
  Round 1 Day 15 | -.33 [-.33 to -.33] | 2.63 [-0.17 to 5.43]
  Round 1 Week 8 | .10 [.10 to .10] | 3.13 [0.40 to 5.87]
  Round 2 Day 5 | -.13 [-.13 to -.13] | 0.68 [0.00 to 1.37]
  Round 2 Day 10: number analyzed (Participants) | 1 | 1
  Round 2 Day 10 | .63 [.63 to .63] | 1.53 [1.53 to 1.53]
  Round 2 Day 15: number analyzed (Participants) | 1 | 1
  Round 2 Day 15 | .47 [.47 to .47] | -0.43 [-0.43 to -0.43]
  Round 2 Week 8: number analyzed (Participants) | 1 | 1
  Round 2 Week 8 | .50 [.50 to .50] | -0.10 [-0.10 to -0.10]

3. Primary Outcome: Change in Upper Extremity Strength - Cylindrical Grip - More Impaired Hand
Description: Change in upper extremity strength compared to baseline assessed using dynamometers to measure grip forces.
Time Frame: Once each intervention week (days 5, 10, and 15), and once at followup (week 8)
Population: 1 subject from SHAM+TESS First group dropped out after round 2 day 5.
Measure: Mean (Full Range); unit: kg
Arm/Group | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First
Number analyzed (Participants) | 1 | 2
kg
  Round 1 Day 5 | 0 [0 to 0] | 0.98 [0 to 1.97]
  Round 1 Day 10 | 0 [0 to 0] | 0.30 [0.00 to 0.60]
  Round 1 Day 15 | .17 [.17 to .17] | 0.77 [0.00 to 1.53]
  Round 1 Week 8 | 0 [0 to 0] | 2.35 [0.00 to 4.70]
  Round 2 Day 5 | 0 [0 to 0] | -2.28 [-4.57 to 0.00]
  Round 2 Day 10: number analyzed (Participants) | 1 | 1
  Round 2 Day 10 | 0 [0 to 0] | 0.27 [0.27 to 0.27]
  Round 2 Day 15: number analyzed (Participants) | 1 | 1
  Round 2 Day 15 | .17 [.17 to .17] | 2.40 [2.40 to 2.40]
  Round 2 Week 8: number analyzed (Participants) | 1 | 1
  Round 2 Week 8 | 0 [0 to 0] | 1.37 [1.37 to 1.37]

ADVERSE EVENTS:
Time Frame: 199 days
Groups:
- Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round 1; Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round 2: Round 1 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 1 Second Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Round 1 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Washout (1 month)
  Round 2 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 2 Second Intervention (4 days):Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Round 2 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
- Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round1; Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round2: Round 1 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 1 Second Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
  Round 1 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Washout (1 month)
  Round 2 First Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice alone for 45 mins.
  Round 2 Second Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after AIH (15x 1.5 mins bouts of 10% oxygen with 1 min intervals of room air).
  Round 2 Third Intervention (4 days): Participants receive 4 consecutive days of TESS during functional task practice for 45 mins after SHAM (15x 1.5 mins bouts of 21% oxygen with 1 min intervals of room air).
Arm/Group | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round 1 | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round 2 | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round1 | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round2
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round 1 (N=1) | Intermittent Hypoxia (AIH) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round 2 (N=1) | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round1 (N=2) | Intermittent Room Air (SHAM) + Transcutaneous Electrical Spinal Cord Stimulation (TESS) First Round2 (N=2)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT04854057/Prot_SAP_000.pdf